CLINICAL TRIAL: NCT05435235
Title: Dapagliflozin in the Prevention of Post-Coronary Intervention Acute Kidney Injury
Brief Title: Dapagliflozin in the Prevention of Post-Coronary Angioplasty Acute Kidney Injury
Acronym: DAPA-PCI-AKI
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Laboratory UNGAL
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Gregg Pressman, Staff Cardiologist and Director of Academics, Cardiology, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022-864
Record Dates: First submitted 2022-06-23; First posted 2022-06-28 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-01

CONDITIONS: Acute Kidney Injury; Percutaneous Coronary Intervention
Keywords: SGLT2 inhibitor; Dapagliflozin; AKI; PCI; Angiography
MeSH Terms: conditions — Acute Kidney Injury | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dapagliflozin arm (Experimental): Patients who received Dapagliflozin 10 mg daily starting 48h prior to PCI and continuing for 48h post-PCI.
  Interventions: Drug: Dapagliflozin 10mg Tab
- Standard of care (No Intervention): Patients who received the standard of care.

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — One tablet daily starting 48h prior to PCI and continuing for 48h post-PCI.
  Arms: Dapagliflozin arm

SUMMARY:
To compare the incidence of acute kidney injury (AKI) post percutaneous coronary intervention (PCI) in a Dapagliflozin treated group versus a group managed with the usual standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or more.
2. Scheduled/non-emergent Percutaneous coronary intervention (PCI).
3. Post-index procedure Staged PCI with at least 14 days from contrast exposure.
4. Patient can fully understand the study information and sign informed consent.

Exclusion Criteria:

1. Cardiogenic shock /need for inotrope or mechanical pump support.
2. Acute kidney injury as defined by KDIGO criteria (<4 weeks) prior to PCI.
3. End-Stage Renal Disease prior to PCI (On renal replacement therapy).
4. Diabetes Mellitus type 1.
5. Active diabetic ketoacidosis or uncontrolled hyperglycemia (blood glucose >400 mg/dl).
6. ST-segment elevation Myocardial Infarction undergoing index PCI.
7. Active Genitourinary infection.
8. Diagnostic Left Heart Catheterization without PCI.
9. Patients undergoing zero contrast PCI.
10. Participation in a randomized controlled pharmaceutical or treatment-related cardiac or pulmonary clinical study within 1 month prior to randomization.
11. Coexistent hemodynamically significant valvulopathy (Symptomatic and/or severe).
12. Patients with Acute Heart Failure admission < 30 days prior to PCI.
13. Intercurrent illness resulting in volume depletion and hypotension (MAP<60 mmHg).
14. Patients with a kidney transplant.
15. Any contrast exposure within 14 days.
16. Patients with estimated glomerular filtration rate (eGFR) < 25 cc/min (Recommended eGFR threshold by Food and Drug Administration labeling).
17. Patients with an active intrinsic inflammatory or autoimmune renal pathology.
18. Women of child bearing age (<50 years old).
19. Prison Inmates

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury | Within 7 days.
  According to the Kidney Disease Improving Global Outcomes (KDIGO) 2012 definition: increase in serum creatinine by ≥ 0.3 mg/dl (≥ 26.5 μmol/l) within 48 hours or increase in serum creatinine (SCr) to ≥ 1.5 times the known baseline which is known or presumed to have occurred within the prior 7 days.
  We will measure Urine Neutrophil Gelatinase-associated Lipocalin (UNGAL) at least 6 hours post-PCI and Serum Creatinine at follow up within 7 days.

SECONDARY OUTCOMES:
Length of hospital stay | 7 days
  Days
Incidence of genitourinary infections | 7 days
  Symptomatic pyuria or new vaginal infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Einstein Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No